CLINICAL TRIAL: NCT05084898
Title: Do Far-UVC Light Devices Reduce the Incidence of Respiratory Viral Illness in Long-term Care Facilities?
Brief Title: Preventing Respiratory Viral Illness Invisibly
Acronym: PRiVII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kenneth Rockwood (Other)
Collaborators: Department of Health, Nova Scotia (Other); Research Nova Scotia (Unknown); Nova Scotia Health Authority (Other)
Responsible Party: Sponsor-Investigator, Kenneth Rockwood, Geriatrician, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 32906-UVC
Record Dates: First submitted 2021-01-26; First posted 2021-10-20 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: COVID-19 Respiratory Infection; Respiratory Virus Infection; Influenza -Like Illness
Keywords: Far-UVC; long-term care; respiratory illnesses; disinfection methods; viral infections
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Intervention Model Description: Residents of three LTC facilities, will be cluster-randomized based on the 'neighbourhoods' they live in (social groups of 18-36) with a 1:1 allocation ratio. Randomization will be stratified by the LTC facility.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: BIinding in this study involves the use of a placebo arm. The placebo lamps will look exactly like the active far-UVC lamps, but they will produce regular fluorescent light and have no disinfection properties.
  The trial will be blinded to everyone involved in the study except for one member of the lead coordinating team who must remain unblinded to provide lamp allocation guidance to the installing electricians. This person will not be involved in data collection or analysis, nor will they have access to participant identifying information, only their deidentified study ID.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Far-UVC light as an additional method of disinfection
  Interventions: Other: Far-UVC light as an additional method of disinfection
- Placebo (Placebo Comparator): "Inactive" fluorescent light (no additional disinfection)
  Interventions: Other: Placebo fluorescent light

INTERVENTIONS:
Other: Far-UVC light as an additional method of disinfection — Far-UVC light is a form of ultraviolet light with an extremely short wavelength (222 nm)
  Arms: Intervention
Other: Placebo fluorescent light — "Inactive" fluorescent light (no additional disinfection)
  Arms: Placebo

SUMMARY:
Elderly people who have multiple health problems are at higher risk of illness from viral respiratory infections, such as influenza (the flu) and COVID-19. This is especially true for residents in long-term care because the usual methods of infection control (handwashing, mask-wearing, and distancing) are difficult to enforce due to the memory problems of many residents and the frequently shared common spaces. It can also be difficult to prevent the spread of viral infections within long-term care because many residents are unable to tell their caregivers when they are feeling ill. Also, some elderly people do not show typical symptoms of infection (like fever), instead they may suddenly become confused or weak.

This study will test if a safe form of ultraviolet light (far-UVC) can be effective as an extra method of disinfection (in addition to usual manual cleaning) against airborne and surface viruses that can cause respiratory infections.

DETAILED DESCRIPTION:
Background: Nova Scotia has the highest proportion of seniors in Canada. Investing in high quality and safe long-term care homes is considered an important healthy aging strategy both here and globally. COVID-19 has disproportionately affected the elderly population, especially those with underlying health conditions. Residents of long-term care (LTC) facilities have been particularly vulnerable during this pandemic in Canada and elsewhere. Several approaches have been mandated to mitigate the high transmissibility of the aerosolised SARS-CoV-2 coronavirus. These are guided by three key principles: minimize time of exposure, maximize distance from sources of virus and finally to shield self from virus. As demonstrated in emerging evidence, these can be effective measures provided ability for compliance and human behaviours. Following life-saving public health guidelines has proven monumentally challenging in LTC facilities, due to the high prevalence of dementia and frailty. These severe public health measures and common infection control measures have resulted in other negative consequences for LTC residents, such as an increased feeling of loneliness, depression, and mental illnesses.

A further challenge with this population is early recognition of RVI in LTC residents can be difficult due to non-specific symptoms and the possibility of atypical presentation and lack of fever in the elderly with influenza. In this population, RVI can present as sudden, unexplained deterioration in physical or mental ability or exacerbation of an underlying condition with no other known cause. Additionally, other underlying conditions could impair residents' abilities to verbalize their symptoms. This could result in delays to the implementation of control and treatment strategies.

Rational: Far-UVC is emerging as a safe form of ultraviolet light disinfectant to kill airborne viral transmissions, including SARS CoV-2 virus. Far-UVC light (207-222 nm) in low doses effectively kills pathogens without damaging exposed human tissues. Preliminary data suggests using the regulatory safe level of exposure of lower dose UVC light (far-UVC light) can inactivate >95% of aerosolized H1N1 influenza virus and 90 percent of human coronaviruses in 8 minutes and almost 100 percent in 25 minutes. Despite growing evidence on far-UVC as a safe and viable infection control strategy, there is limited research on the feasibility, acceptability and efficacy of far-UVC in LTC settings.

Main Objective: To determine whether far-UVC light causes a reduction in the incidence of influenza-like illnesses, respiratory infections, and COVID-19 infections, among residents in long term care facilities.

Methodology: This is a cluster randomized control trial designed to identify superiority of the intervention. Residents of three LTC facilities, will be cluster-randomized based on the 'neighbourhoods' they live in (social groups of 18-36) with a 1:1 allocation ratio. Randomization will be stratified by the LTC facility. Neighbourhoods will be randomly assigned to have either 222 nm far-UVC lights installed in common areas (treated) or matching placebo lights without far-UVC capabilities (control). Both groups will still receive standard disinfecting procedures and are subject to Nova Scotia's COVID prevention measures. The far-UVC and fluorescent lights will be placed in high traffic areas (e.g. dining rooms, main corridors). Residents spend approximately 3-4 hours daily in these common areas. The far-UVC lamps will be kept at a wavelength of 222 nm and exposure times that have been demonstrated to be safe for use among elderly populations. The trial period will span over 2-3 flu seasons to allow for sufficient data and sample size to describe the efficacy and sustainability of the far-UVC intervention. To be responsive to key policy and planning needs during post pandemic times, findings will be presented routinely to advisory council members and to relevant stakeholders in the province.

ELIGIBILITY:
Exclusion Criteria: LTC residents who do not consent to data collection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
A diagnosis of COVID-19 or other respiratory viral infection | Over 3 flu seasons, approximately 28 months
  Diagnosis will be based on positive laboratory finding of SARS-CoV-2, influenza A, influenza B, respiratory syncytial virus, or other respiratory viral infections (as per available testing). Testing will be performed on nasal swabs collected from participants who are positive for any of the symptoms in the screening protocol.

SECONDARY OUTCOMES:
Time to recovery or death | From the date of diagnosis until the date of recovery or date of death, whichever comes first, assessed up to 30 days.
  Number of days from diagnosis of respiratory viral infection until recovery or death. Participant will be deemed "recovered" once their overall health status (vital, functional, and cognitive) has been stable for one week. This return to stable state will be determined by participant's clinical care team and is part of usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Rockwood, MD, Principal Investigator — Nova Scotia Health Authority
Locations (3):
- Canada (3):
  - Northwood Halifax Campus, Halifax, Nova Scotia
  - The Cove Guest Home, Sydney, Nova Scotia
  - Windsor Elms Village, Windsor, Nova Scotia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andrew M, Searle SD, McElhaney JE, McNeil SA, Clarke B, Rockwood K, Kelvin DJ. COVID-19, frailty and long-term care: Implications for policy and practice. J Infect Dev Ctries. 2020 May 31;14(5):428-432. doi: 10.3855/jidc.13003. PMID 32525825
- [Background] Austin PC. A Tutorial on Multilevel Survival Analysis: Methods, Models and Applications. Int Stat Rev. 2017 Aug;85(2):185-203. doi: 10.1111/insr.12214. Epub 2017 Mar 24. PMID 29307954
- [Background] Buonanno M, Welch D, Shuryak I, Brenner DJ. Far-UVC light (222 nm) efficiently and safely inactivates airborne human coronaviruses. Sci Rep. 2020 Jun 24;10(1):10285. doi: 10.1038/s41598-020-67211-2. PMID 32581288
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Garner R, Tanuseputro P, Manuel DG, Sanmartin C. Transitions to long-term and residential care among older Canadians. Health Rep. 2018 May 16;29(5):13-23. PMID 29852053
- [Background] Moberg J, Kramer M. A brief history of the cluster randomised trial design. J R Soc Med. 2015 May;108(5):192-8. doi: 10.1177/0141076815582303. No abstract available. PMID 26022551
- [Background] Pallmann P, Bedding AW, Choodari-Oskooei B, Dimairo M, Flight L, Hampson LV, Holmes J, Mander AP, Odondi L, Sydes MR, Villar SS, Wason JMS, Weir CJ, Wheeler GM, Yap C, Jaki T. Adaptive designs in clinical trials: why use them, and how to run and report them. BMC Med. 2018 Feb 28;16(1):29. doi: 10.1186/s12916-018-1017-7. PMID 29490655
- [Background] Welch D, Buonanno M, Grilj V, Shuryak I, Crickmore C, Bigelow AW, Randers-Pehrson G, Johnson GW, Brenner DJ. Far-UVC light: A new tool to control the spread of airborne-mediated microbial diseases. Sci Rep. 2018 Feb 9;8(1):2752. doi: 10.1038/s41598-018-21058-w. PMID 29426899
- [Background] Kirk MA, Kelley C, Yankey N, Birken SA, Abadie B, Damschroder L. A systematic review of the use of the Consolidated Framework for Implementation Research. Implement Sci. 2016 May 17;11:72. doi: 10.1186/s13012-016-0437-z. PMID 27189233
- [Background] Liu K, Chen Y, Lin R, Han K. Clinical features of COVID-19 in elderly patients: A comparison with young and middle-aged patients. J Infect. 2020 Jun;80(6):e14-e18. doi: 10.1016/j.jinf.2020.03.005. Epub 2020 Mar 27. PMID 32171866
- [Background] Liu Y, Mao B, Liang S, Yang JW, Lu HW, Chai YH, Wang L, Zhang L, Li QH, Zhao L, He Y, Gu XL, Ji XB, Li L, Jie ZJ, Li Q, Li XY, Lu HZ, Zhang WH, Song YL, Qu JM, Xu JF; Shanghai Clinical Treatment Experts Group for COVID-19. Association between age and clinical characteristics and outcomes of COVID-19. Eur Respir J. 2020 May 27;55(5):2001112. doi: 10.1183/13993003.01112-2020. Print 2020 May. PMID 32312864
- [Background] Armitage R, Nellums LB. COVID-19 and the consequences of isolating the elderly. Lancet Public Health. 2020 May;5(5):e256. doi: 10.1016/S2468-2667(20)30061-X. Epub 2020 Mar 20. No abstract available. PMID 32199471
- [Background] Simard J, Volicer L. Loneliness and Isolation in Long-term Care and the COVID-19 Pandemic. J Am Med Dir Assoc. 2020 Jul;21(7):966-967. doi: 10.1016/j.jamda.2020.05.006. Epub 2020 May 8. No abstract available. PMID 32505516
- [Background] El Haj M, Altintas E, Chapelet G, Kapogiannis D, Gallouj K. High depression and anxiety in people with Alzheimer's disease living in retirement homes during the covid-19 crisis. Psychiatry Res. 2020 Sep;291:113294. doi: 10.1016/j.psychres.2020.113294. Epub 2020 Jul 13. PMID 32763552
- [Background] Falsey AR, Baran A, Walsh EE. Should clinical case definitions of influenza in hospitalized older adults include fever? Influenza Other Respir Viruses. 2015 Aug;9 Suppl 1(Suppl 1):23-9. doi: 10.1111/irv.12316. PMID 26256292
- [Background] Sayers G, Igoe D, Carr M, Cosgrave M, Duffy M, Crowley B, O'Herlihy B. High morbidity and mortality associated with an outbreak of influenza A(H3N2) in a psycho-geriatric facility. Epidemiol Infect. 2013 Feb;141(2):357-65. doi: 10.1017/S0950268812000659. Epub 2012 Apr 17. PMID 22672856
- [Background] Drinka PJ, Krause P, Nest L, Gravenstein S, Goodman B, Shult P. Delays in the application of outbreak control prophylaxis for influenza A in a nursing home. Infect Control Hosp Epidemiol. 2002 Oct;23(10):600-3. doi: 10.1086/501978. PMID 12400890
- [Background] Mahmud SM, Thompson LH, Nowicki DL, Plourde PJ. Outbreaks of influenza-like illness in long-term care facilities in Winnipeg, Canada. Influenza Other Respir Viruses. 2013 Nov;7(6):1055-61. doi: 10.1111/irv.12052. Epub 2012 Nov 12. PMID 23145997
- [Derived] Nix HP, Meeker S, King CE, Andrew M, Davis IRC, Koto PS, Sim M, Murdoch J, Patriquin G, Theriault C, Reidy S, Rockwood M, Sampalli T, Searle SD, Rockwood K. Preventing Respiratory Viral Illness Invisibly (PRiVII): protocol for a pragmatic cluster randomized trial evaluating far-UVC light devices in long-term care facilities to reduce infections. Trials. 2024 Jan 26;25(1):88. doi: 10.1186/s13063-024-07909-0. PMID 38279184